CLINICAL TRIAL: NCT04821024
Title: Evaluation of the Relationship Between Neck Pain and Ergonomic Factors in Office Workers
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021/18
Record Dates: First submitted 2021-03-26; First posted 2021-03-29 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Disability Physical; Neck Pain; Ergonomic Factors
Keywords: neck pain office workers ergonomic factors
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mild-moderate disability: Those whose neck disability index value is 5-34
  Interventions: Diagnostic Test: A self-administered questionnaire
- high disability: Those whose neck disability index value is 35 and above
  Interventions: Diagnostic Test: A self-administered questionnaire

INTERVENTIONS:
Diagnostic Test: A self-administered questionnaire — A self-administered questionnaire will be used to screen Neck disability index, demographic information and ergonomic risk factors.

SUMMARY:
The current study aimed to explore the associations between disability levels and occupational risk factors in computer-using office workers with neck pain.

DETAILED DESCRIPTION:
This is a cross-sectional study. All participants will provide informed consent before participating in the study. The study will be conducted in accordance with the Helsinki Declaration criteria. Data will be collected using questionnaires, which include information on demographic, clinical, and occupational ergonomic conditions.

Patients will be divided into 2 groups as mild-moderate and severe disabled according to their neck disability index values and will be analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 55,
* working on computer,
* having neck pain at least three months.

Exclusion Criteria:

* reporting pregnancy,
* having a history of accidents,
* trauma or surgery in the neck region,
* congenital anomaly of the spine,
* rheumatologic disease,
* osteoporosis,
* spondylosis,
* spondylolisthesis,
* infection of the spine
* cervical disc herniation,
* tumor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: aged between 18 and 55, working on computer, having neck pain at least three months
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
neck disability index | 1 interview day
  The Neck Disability Index (NDI) is a self-report questionnaire used to determine how neck pain affects a patient's daily life and to assess the self-rated disability of patients with neck pain
Rapid Office Strain Assessment | 1 interview day
  Rapid Office Strain Assessment is a method that determined the potential ergonomic risk factors computer position, computer screen position, head, and back position, and mouse position.

CONTACTS AND LOCATIONS:
Overall Officials: cansın medin-ceylan, MD, Principal Investigator — istanbul physical medicine rehabilitation research and training hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Research and Training Hospital, Istanbul, Bahçelievler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cote P, van der Velde G, Cassidy JD, Carroll LJ, Hogg-Johnson S, Holm LW, Carragee EJ, Haldeman S, Nordin M, Hurwitz EL, Guzman J, Peloso PM; Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. The burden and determinants of neck pain in workers: results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Spine (Phila Pa 1976). 2008 Feb 15;33(4 Suppl):S60-74. doi: 10.1097/BRS.0b013e3181643ee4. PMID 18204402
- [Background] Aas RW, Tuntland H, Holte KA, Roe C, Lund T, Marklund S, Moller A. Workplace interventions for neck pain in workers. Cochrane Database Syst Rev. 2011 Apr 13;2011(4):CD008160. doi: 10.1002/14651858.CD008160.pub2. PMID 21491405
- [Background] Vassilaki M, Hurwitz EL. Insights in public health: perspectives on pain in the low back and neck: global burden, epidemiology, and management. Hawaii J Med Public Health. 2014 Apr;73(4):122-6. No abstract available. PMID 24765562
- [Background] Matsudaira K, Kawaguchi M, Isomura T, Inuzuka K, Koga T, Miyoshi K, Konishi H. Assessment of psychosocial risk factors for the development of non-specific chronic disabling low back pain in Japanese workers-findings from the Japan Epidemiological Research of Occupation-related Back Pain (JOB) study. Ind Health. 2015;53(4):368-77. doi: 10.2486/indhealth.2014-0260. Epub 2015 Jun 6. PMID 26051289
- [Background] McLean SM, May S, Klaber-Moffett J, Sharp DM, Gardiner E. Risk factors for the onset of non-specific neck pain: a systematic review. J Epidemiol Community Health. 2010 Jul;64(7):565-72. doi: 10.1136/jech.2009.090720. Epub 2010 May 12. PMID 20466711
- [Derived] Medin-Ceylan C, Korkmaz MD, Sahbaz T, Cigdem Karacay B. Risk factors of neck disability in computer-using office workers: a cross-sectional study. Int J Occup Saf Ergon. 2023 Mar;29(1):44-49. doi: 10.1080/10803548.2021.2021712. Epub 2022 Feb 6. PMID 34952560